CLINICAL TRIAL: NCT02578953
Title: Bioequivalence Study of Dutasteride Capsules-An Evaluation of the Bioequivalence of Dutasteride Capsule Manufactured at GSK Compared to Dutasteride Capsule Manufactured at Catalent in Healthy Japanese Male Subjects
Brief Title: Bioequivalence Study of Dutasteride Capsules in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204646
Record Dates: First submitted 2015-09-10; First posted 2015-10-19 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: Bioequivalence; Fasted state; Japanese male healthy subjects; Dutasteride
MeSH Terms: conditions — Prostatic Hyperplasia; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1-Dutasteride test product and then Reference product (Experimental): Participants will receive treatment A in period 1 and treatment B in period 2. Where treatment A= dutasteride 0.5 mg capsule test product, treatment B= dutasteride 0.5 mg capsule reference product.
  Interventions: Drug: Dutasteride-Test product; Drug: Dutasteride-Reference product
- Sequence 2-Dutasteride reference product and then test product (Experimental): Participants will receive treatment B in period 1 and treatment A in period 2. Where treatment A= dutasteride 0.5 mg capsule test product, treatment B= dutasteride 0.5 mg capsule reference product.
  Interventions: Drug: Dutasteride-Test product; Drug: Dutasteride-Reference product

INTERVENTIONS:
Drug: Dutasteride-Test product — Dutasteride Capsules are oblong, opaque, dull-yellow, gelatin capsules. The capsules contain 0.5 mg dutasteride for oral administration. The capsules also contain Butylated Hydroxytoluene, Mono-di-glycerides of Caprylic/Capric Acid (MDC), Gelatin, Concentrated Glycerin, Titanium Dioxide, Iron Oxide Yellow as ingredients. This product will be manufactured by GSK, Poznan.
Drug: Dutasteride-Reference product — Dutasteride Capsules are oblong, opaque, dull-yellow, gelatin capsules. The capsules contain 0.5 mg dutasteride for oral administration. The capsules also contain Butylated Hydroxytoluene, Mono-di-glycerides of Caprylic/Capric Acid (MDC), Gelatin, Glycerin, Concentrated Glycerin, Titanium Dioxide, Iron Oxide Yellow as ingredients. This product will be manufactured by Catalent, Beinheim.

SUMMARY:
This will be a single center, open-label, single dose, randomized and 2-way crossover study in healthy Japanese male subjects under fasting conditions. The study will be conducted to determine the bioequivalence between dutasteride capsules manufactured at GSK (test product) and dutasteride capsule manufactured at Catalent (reference product) in healthy Japanese male subjects. Subjects will have a screening visit within 30 days prior to the first dose of study treatment, two treatment periods separated by 28-days washout period, a re-visit 10-14 days after the second dose for the first follow-up and a second follow up via telephone 50-54 days after the second dose. The total duration of the study will be approximately 15 weeks from screening to the second follow up.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 64 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18.5-24.9 kg/meter squared at screening.
* Japanese male.
* Male subjects with female partners of child bearing potential must comply with the contraception requirements from the time of first dose of study medication until the second follow-up.
* Capable of giving signed informed consent as described in which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* ALT and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT interval (QTc) >450 milliseconds (msec).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident.
* History of diabetes or peptic ulcer disease which is uncontrolled by medical management.
* History of breast cancer or clinical breast examination finding suggestive of malignancy.
* History of malignancy within the past five years, except for basal cell carcinoma of the skin. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* Prior medical history or evidence of prostate cancer (e.g., positive biopsy, or suspicious ultrasound, or suspicious digital rectal examination (DRE)). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study.
* Creatinine >1.5xULN.
* History or current conditions of drug abuse or alcoholism.
* Unable to refrain from the use of prescription drugs, non- prescription drugs, vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks. One drink is equivalent to 350 milliliter (mL) of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy.
* The subject is positive Serological test for syphilis (Rapid plasma reagin test and Treponema pallidum), Human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HbsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening.
* A positive pre-study drug screen.
* Where participation in the study would result in donation of blood or blood products >=400 mL within 4 months or >=200 mL within 1 month.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within 4 months prior to the first dosing day in the current study.
* The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC 0-t) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Maximal measured plasma concentration (Cmax) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.

SECONDARY OUTCOMES:
Number of subjects with adverse events | Approximately 12 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Change from Baseline in hematology parameters | Baseline (screening or Day-1) and Day 2 of each treatment period.
  Hematology parameters includes: red blood cells (RBC) count, white blood cell (WBC) count (absolute), platelet count, hemoglobin, hematocrit, RBC indices (mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration)
Change from Baseline in clinical chemistry parameters | Baseline (screening or Day-1) and Day 2 of each treatment period.
  Clinical chemistry parameters includes: blood urea nitrogen, creatinine, uric acid, creatin phosphokinase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase, alkarine phosphatise (ALP), amylase, lactate dehydrogenase, total and direct bilirubin, albumin, fasting glucose, total protein, triglyceride, total cholesterol, high density lipoprotein -cholesterol, low density lipoprotein -cholesterol, potassium, chloride, calcium, phosphorus and sodium.
Change from Baseline in routine urinalysis parameters | Baseline (screening or Day-1) and Day 2 of each treatment period.
  Routine urinalysis parameters includes: Specific gravity; pH, glucose, protein, blood and ketones, bilirubin and urobilinogen by dipstick; Sediment.
Change from Baseline in systolic and diastolic blood pressure measurements | Baseline (screening) and Day 1and Day 2 of each treatment period and at first follow-up visit (approximately up to 11 weeks).
  Blood pressure measurements will be collected at screening; pre-dose and 3 hours, 24 hours post-dose in each period; and first follow-up visit.
Change from Baseline in pulse rate | Baseline (screening) and Day 1and Day 2 of each treatment period and at first follow-up visit (approximately up to 11 weeks).
  Pulse rate measurement will be collected at screening; pre-dose and 3 hours, 24 hours post-dose in each period; and first follow-up visit.
Change from Baseline in electrocardiogram (ECG) parameters | Baseline (screening) and Day 1and Day 2 of each treatment period and at first follow-up visit (approximately up to 11 weeks).
  Electrocardiograms (ECGs) will be recorded whilst the subject is in a supine position, after 10 minutes of rest. Baseline will be defined as the mean of the three pre-dose measurements (separated by a minimum of 5 minutes) that occurred pre-dose on Day 1.
Change from Baseline in body temperature | Baseline (screening) and Day 1and Day 2 of each treatment period and at first follow-up visit (approximately up to 11 weeks).
  Body temperature measurement will be collected at screening; pre-dose and 3 hours, 24 hours post-dose in each period; and first follow-up visit.
Area under the concentration-time curve from pre-dose to 24 hours (AUC[0-24]) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Area under the plasma concentration-time curve from time zero to infinity (AUC 0-infinity) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Time of the maximum plasma concentration (tmax) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Elimination rate constant (Kel) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Terminal half life (t1/2e) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Percentage of AUC0-infinity obtained by extrapolation (%AUCex) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Apparent clearance following oral dosing (CL/F) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Apparent volume of distribution after oral administration (Vz/F) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Mean residence time (MRT) of dutasteride test product and reference product | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.
Correlation coefficient between time and log concentration of dutasteride for the points used in the estimation of kel. | Pre-dose and at the following times post dose: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours) in each period.
  Blood samples will be collected for PK analyses in each period before dosing (0 hour) and at the following times after the dose 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 6, 8, 10, 12, 18, 24, 36, 48 and 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 204646 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/204646?search=study&b'study_ids=204646'#rs
- Available data/document: Statistical Analysis Plan: 204646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 204646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 204646 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register